CLINICAL TRIAL: NCT01549795
Title: Trapianto di Fegato Per Colangiocarcinoma (CCA) Ilare in Associazione a Radio e Chemioterapia Neoadiuvante
Brief Title: Liver Transplantation for Hilar Cholangiocarcinoma in Association With Neoadjuvant Radio- and Chemo-therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Director of the Hepatobiliary Surgery and Liver Transplantation Unit, Azienda Ospedaliera di Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2372P
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Hilar Cholangiocarcinoma; Primary Sclerosing Cholangitis
Keywords: Liver transplantation; Neoadjuvant radio- chemo-therapy
MeSH Terms: conditions — Klatskin Tumor; Cholangitis, Sclerosing | interventions — Liver Transplantation; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Liver transplantation — Liver transplantation using classic technique and avoiding proximal ilum dissection. The donor hepatic artery will be anastomosed to a jump graft connected to the Aorta. In case of positive margin of the bile duct at a frozen section analysis the liver transplant will be performed after an adjunctive pancreatodudodenctomy
Radiation: 45 Gy external radiations — 45 Gy in 30 fractions, 1,5 Gy twice a day) and 5-FU iv infusion- 3 week treatment
Radiation: Endoluminal bile duct Brachytherapy — Brachytherapy (20 Gy a 1 cm in 20-25h) - administered 2 weeks after radiotherapy completion
Drug: Capecitabine — Capecitabine - administered till liver transplantation
Procedure: Pre liver transplantation laparoscopic hand assisted staging — Pre liver transplantation laparoscopic hand assisted staging for sampling hepatic artery lymph nodes and assessing peritoneal disease.

SUMMARY:
Single-arm pilot clinical trial. Patients with non operable CC associated with PSC will be subjected to liver transplantation after a neoadjuvant multimodal therapy protocol.

Cholangiocarcinoma (CC) accounts for 3% of all gastrointestinal cancers; it is more frequent in patients with primary sclerosing cholangitis (PSC), who carry an 8%-12% risk of developing this type of neoplasm. Only a minority of patients are suitable for resection partly because of the anatomic position of the tumor (which often arises from the bile duct bifurcation) and partly because of the frequently coexisting liver disease. In fact, CC is currently considered a major contraindication to liver transplantation (OLT) at the majority of centers, given a 5-year survival rate of 0%-35%.

New strategies have been developed for the treatment of this kind of cancer arising in PSC. The Nebraska University group showed a 1 and 3 years survival of 55 and 45 % combining a neoadjuvant intra bile duct barchytherapy and 5-FU based chemotherapy with liver transplantation. University of Pittsburg proposed also a neoadjuvant protocol prior to liver transplantation based on systemic chemotherapy and external radiotherapy reporting a 53% 5 years survival. More convincing results come from the Mayo Clinic. An accurate selection of patients and a proper neoadjuvant multimodal therapy (chemotherapy, external radiotherapy and intraluminal bile duct brachytherapy) lead to a 80% 5 years survival after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Male or female
* Diagnosis of Cholangiocarcinoma using:
* PTBD biopsy or Brushing cytology
* Ca 19-9>100mg/ml and/or liver mass at CT or MRI with malignant stenosis apperance at Cholangiography,
* Non resectable tumour araising above the cystic duct
* Absence of intra and extra hepatic metastasis
* ECOG score(Eastern Cooperative Oncology Group) 0
* ASA score (American Society of Anesthesiologists) ≤ 3
* Ability to understand and willingness to sign the written informed consent form (ICF)

Exclusion Criteria:

* Intrahepatic Cholangiocarcinoma
* Non controlled infection
* Previous radio or chemotherapy
* Previsous bile duct resection or attempt to resection
* Intra and/or extrahepatic metastasis
* Preivious malignant neoplasm (within 5 years)
* Execution of trans peritoneal biopsy
* Tumour diameter more than 3 cm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients free of disease at 24 months post-transplant | 24 months
Time to recurrence after liver transplant | 24 months

SECONDARY OUTCOMES:
Progression disease free survival | 24 months
Overall 2 years survival after liver transplantation | 24 months
Complication rate due to radiotherapy (Hepatic artery thrombosis and Portal vein thrombosis) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Cillo, MD, Study Chair — Azienda Ospedaliera di Padova; Enrico Gringeri, MD, Principal Investigator — Azienda Ospedaliera di Padova
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Padova, Italy

REFERENCES:
- [Background] Hemming AW, Reed AI, Fujita S, Foley DP, Howard RJ. Surgical management of hilar cholangiocarcinoma. Ann Surg. 2005 May;241(5):693-9; discussion 699-702. doi: 10.1097/01.sla.0000160701.38945.82. PMID 15849505
- [Background] Rea DJ, Heimbach JK, Rosen CB, Haddock MG, Alberts SR, Kremers WK, Gores GJ, Nagorney DM. Liver transplantation with neoadjuvant chemoradiation is more effective than resection for hilar cholangiocarcinoma. Ann Surg. 2005 Sep;242(3):451-8; discussion 458-61. doi: 10.1097/01.sla.0000179678.13285.fa. PMID 16135931
- [Background] Rosen CB, Heimbach JK, Gores GJ. Liver transplantation for cholangiocarcinoma. Transpl Int. 2010 Jul;23(7):692-7. doi: 10.1111/j.1432-2277.2010.01108.x. Epub 2010 May 20. PMID 20497401
- [Background] Hamilton JP. Epigenetic mechanisms involved in the pathogenesis of hepatobiliary malignancies. Epigenomics. 2010 Apr 1;2(2):233-243. doi: 10.2217/epi.10.9. PMID 20556199
- See also: Hepatobiliary surgery and Liver Transplantation Unit, University Hospital of Padua (Italy) — http://www.fegatochirurgia.com